CLINICAL TRIAL: NCT04168619
Title: Methotrexate-related Liver Toxicity in Psoriasis Patients, Using Ultrasound-based Techniques as a Diagnostic Tool
Brief Title: MTX-related Liver Toxicity in Psoriasis Patients, Using Ultrasound-based Techniques as a Diagnostic Tool
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Sze-Man Wong, Honorary Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 19-390
Record Dates: First submitted 2019-10-25; First posted 2019-11-19 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis; Liver Fibrosis
Keywords: Liver Fibrosis; Psoriasis; Methotrexate; Transient elastography; Two-dimensional shear wave elastrography
MeSH Terms: conditions — Psoriasis; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transient elastography (TE): All patients who had MTX taken
  Interventions: Drug: Discontinue methotrexate
- Two dimensional shear wave elastography (2D SWE): For patients who has cumulative more than 3.5g methotrexate
  Interventions: Drug: Discontinue methotrexate
- Liver biopsy: For patients who has cumulative more than 3.5g methotrexate and had 2D SWE done
  Interventions: Drug: Discontinue methotrexate; Other: Medication depends on clinical judgement

INTERVENTIONS:
Drug: Discontinue methotrexate — According to the international guideline, patients with Roenigk grade 3a which indicate methotrexate-induced liver injury may continue methotrexate with a repeat biopsy in 6 months. In patients with Roenigk grades 3b or 4, indicate significant liver fibrosis/cirrhosis, methotrexate should be discontinued.
Other: Medication depends on clinical judgement — Once discontinued methotrexate, based on subject's clinical condition and prescribe alternative treatment
  Groups: Liver biopsy

SUMMARY:
Methotrexate is one of the commonly used conventional systemic treatment for moderate to severe psoriasis as well as psoriatic arthritis. It is also used as co-therapy with TNF-antagonists to improve efficacy and reduce neutralizing drug antibodies formation. Apart from the bone marrow suppression, which can largely be avoided with careful dosing, monitoring and avoidance of certain drug interaction, hepatotoxicity is one of the major side-effects. The prevalence of significant liver fibrosis in patients taking methotrexate is estimated to be 5% and cirrhosis 1-2%.

The British Association of Dermatologist's guideline (2016) discussed a few non-invasive tests such as the amino-terminal peptide of procollagen III (PIIINP), Fibrotest and transient elastography. While PIIINP was recommended to be used in baseline and serial assessment, liver stiffness measurement by transient elastography is not yet widely used owing to lack of high-quality data. Transient elastography (TE) has been shown to correlate well with liver fibrosis and has been widely adopted as a non-invasive method to assess liver fibrosis in various chronic liver disease.

Two-dimensional shear wave elastrography (2D SWE) is a novel ultrasound technique that combines shear wave elastography with traditional ultrasound imaging. Liver stiffness measurement can be performed under the guidance of high rate B-mode image, allowing real-time visualization of liver parenchyma and avoidance of non-target structures such as vessels or focal liver lesions.

In view of the demand of a safer and reliable non-invasive test to detect advanced liver fibrosis in psoriasis patients receiving methotrexate, we propose to recruit at-risk patients for a paired TE and 2D SWE assessment and liver biopsy.

DETAILED DESCRIPTION:
Methotrexate is one of the commonly used conventional systemic treatment for moderate to severe psoriasis as well as psoriatic arthritis. It is also used as co-therapy with TNF-antagonists to improve efficacy and reduce neutralizing drug antibodies formation. Apart from the bone marrow suppression, which can largely be avoided with careful dosing, monitoring and avoidance of certain drug interaction, hepatotoxicity is one of the major side-effects. Short term rises in hepatic transaminases are well recognized with methotrexate, which is largely reversible. However, the insidious development of liver fibrosis and ultimately cirrhosis is of greater clinical concern given this may be irreversible with significant impact. Methotrexate-induced liver fibrosis is still a concern especially in patients who received high cumulative dose and those with comorbid risk factors such as diabetes and obesity. The prevalence of significant fibrosis and cirrhosis were reported to be 4.5 - 33.3% and 0 - 25.6%, respectively, in liver biopsy series of psoriasis patients on methotrexate. The results were so variable owing to the facts that many studies were old with poor reporting and variable histological scoring system making interpretation difficult.

According to the NICE guideline and British Association of Dermatologist's guideline ( 2016), liver biopsy remains the gold standard in the assessment of liver fibrosis, however, it is a relatively invasive procedure, with potential sampling error and inter-observer variability, leading to decreasing use of liver biopsy as routine for monitoring methotrexate hepatotoxicity . Non-invasive methods to assess liver fibrosis are therefore advocated, including serum indices as well as transient elastography.

Transient elastography has been shown to correlate well with liver fibrosis in chronic hepatitis and has been widely adopted as a noninvasive method to assess liver fibrosis in various chronic liver disease, but not yet in this specific Psoriasis patients on methotrexate. There is increasing trend to use transient elastography for detection of methotrexate-associated liver fibrosis. However, only few studies included adequate number of patients with concomitant liver biopsy and transient elastography. Data from a study including a relatively high number of patients with liver biopsy (24 psoriasis patients) reported successful scan rate of 83.3% and high negative predictive value of 88% for significant fibrosis. Alternative, Serum procollagen III level (PIIINP) for liver fibrosis is only available in selected specialist centres oversea but not in HK and is costly. Currently, psoriasis patients on methotrexate with cumulative dose of 3000mg of above are advised to have USG guided Fine-needle aspiration (FNA) liver biopsy to assess the presence of liver fibrosis with severity grading , according to American Academy of Dermatology Guideline in Methotrexate dosing. For patient with liver fibrosis grading of 3 a or above ( Roenigfk classification) , they are advised to stop methotrexate and switch to alternative medication. In view of the demand of a safer and reliable non-invasive test to detect advanced liver fibrosis in psoriasis patients receiving methotrexate, we propose to recruit these patients for a paired transient elastography assessment and liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis who are managed in the Dermatology or Dermatology-Rheumatology combined Clinic, Queen Mary Hospital, Hong Kong, will be identified. Patients with clinical diagnosis of psoriasis or psoriatic arthropathy treated with ≥ 3.5 grams of methotrexate in the past or currently will be recruited.

Exclusion Criteria:

* Patients with contraindications for liver biopsy e.g. bleeding tendencies
* Patients with known decompensated cirrhosis
* Pregnancy
* Unstable medical illness or active infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of psoriasis or psoriatic arthropathy treated with ≥ 3.5 grams of methotrexate in the past or currently
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate | At the time of diagnostic procedure
  The meanTE value of psoriasis patients detected with liver injury (. Roenigk. Grade 3a) and liver fibrosis Roenigk grade 3b and above) Area under the receiver operating characteristic curve (AUROC) will be performed to assess if TE is capable of identifying patients with and without liver injury
Performance characteristics | At the time of diagnostic procedure
  Area under the receiver operating characteristic curve (AUROC) will be performed to assess if TE and Shear wave elastography( SW). is capable of identifying patients with and without liver injury

SECONDARY OUTCOMES:
Evaluate risk factors of liver fibrosis | At the time of diagnostic procedure
  Subject's demographic information eg age gender, cumulative dose of MTX, duration of disease. Presence of PsA and other comorbidities will be collected and assessed if there is any relationship of methotrexate induce liver injury.
Relationship of cumulative methotrexate dose | At the time of diagnostic procedure
  Use the relationship of cumulative methotrexate dose, TE score and liver biopsy grade to identify the best cut-off value of liver stiffness for advanced liver fibrosis in psoriasis patients on methotrexate

CONTACTS AND LOCATIONS:
Overall Officials: Sze-man Wong, MSc, Principal Investigator — The University of Hong Kong
Locations (1):
- Division of Dermatology, Department of Medicine, Faculty of Medicine, University of Hong Kong, Central, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.